CLINICAL TRIAL: NCT03019575
Title: A Phase III, Multi-Center, Open Label, Single-Group Trial to Investigate the Efficacy and Safety of MK-8962 (Corifollitropin Alfa) in Combination With Human Chorionic Gonadotropin (hCG) for Initiation or Restoration of Puberty as Assessed by Increased Testicular Volume in Adolescent Males 14 to <18 Years Old With Hypogonadotropic Hypogonadism (MK-8962-043)
Brief Title: Efficacy and Safety of Corifollitropin Alfa (MK-8962) in Combination With Human Chorionic Gonadotropin (hCG) in Adolescent Males With Hypogonadotropic Hypogonadism (HH) (MK-8962-043)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8962-043; 2015-001878-18 (EudraCT Number); MK-8962-043 (Other: Merck)
Record Dates: First submitted 2017-01-11; First posted 2017-01-12 (Estimated); Results first posted 2021-04-08 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2022-02

CONDITIONS: Hypogonadotropic Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — follicle stimulating hormone, human, with HCG C-terminal peptide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Corifollitropin alfa (CFA)+human Chorionic Gonadotropin (hCG) (Experimental): Participants received 100 μg (if body weight was ≤60 kg) or 150 μg (if body weight was >60 kg) of CFA as a subcutaneous (SC) injection once every 2 weeks for 64 Weeks (Day 1, Week 0 through Week 64) and 500-5000 IU of hCG reconstituted with 1 ml of 0.9% sodium chloride solution, as a SC injection twice a week for 52 weeks (last day of Week 12 through Week 64). The total treatment duration was 64 Weeks.
  Interventions: Drug: Corifollitropin alfa; Drug: hCG

INTERVENTIONS:
Drug: Corifollitropin alfa — CFA administered 100 μg (if body weight ≤60 kg) or 150 μg (if body weight >60 kg) by SC injection, once every 2 weeks for 64 weeks (Day 1, Week 0 through Week 64).
  Other Names: MK-8962; Elonva
Drug: hCG — hCG 500-5000 IU reconstituted with 1 ml of 0.9% sodium chloride solution, as a SC injection twice a week for 52 weeks (last day of Week 12 through Week 64).

SUMMARY:
The purpose of the study is to investigate whether corifollitropin alfa (MK-8962), administered alone for 12 weeks and then in combination with human chorionic gonadotropin (hCG) for 52 weeks, increases the testicular volume in adolescent males aged 14 to <18. In addition, the study will evaluate participants for safety, tolerability and for the development of corifollitropin alfa antibodies. No formal hypothesis will be tested for this estimation study

ELIGIBILITY:
Inclusion Criteria:

* Have legal representative who understands the study procedures, alternative treatments available and risks involved with the study, and voluntarily agrees to the individual's participation by giving written informed consent, and the individual has an age-appropriate understanding of the same to give informed written assent if applicable.
* Diagnosed with hypogonadotropic hypogonadism (either isolated or associated with panhypopituitarism), either congenital or acquired with onset prior to puberty.
* Have bilateral pre-gonadarche testes as defined by testicular volume <4.0 mL for each testicle, as determined by ultrasound and assessed by the investigator (if qualified) or local radiologist with appropriate training and expertise in reading testicular ultrasound. Note: participants with a volume of <4.0 mL in one testicle and a volume of 4-8 mL in the other testicle are considered to be pre-gonadarche and may participate, if there is no history or evidence of a primary testicular disorder (see Exclusion Criteria 1 and 2).
* Have circulating levels of total testosterone (Total T) less than the lower limit of normal (LLN) of 8.3 nmol/L as specified by the central lab for a young healthy adult male.
* Have follicle stimulating hormone (FSH) ≤2 IU/L and luteinizing hormone (LH) ≤2 IU/L.
* Have inhibin-B levels ≤35 pg/mL. (Note: if individual has inhibin-B levels >35 pg/mL, but meets all of the other inclusion/exclusion criteria, either a GnRH agonist (GnRHa) stimulation test or GnRH IV infusion test may be performed.
* In good general physical and mental health, in the opinion of the investigator/sponsor, as assessed by physical examination and routine clinical laboratory tests.
* Have a parent/guardian able and willing to support the individual's participation by supporting adherence to study drug dosing and visit schedules.

Exclusion Criteria:

* Have a history of bilateral cryptorchidism (maldescended testes) or unilateral cryptorchidism treated after the age of 2 years.
* Have a history or presence of clinically significant testicular problems (e.g., epididymitis, orchitis, testicular torsion, varicocele Grade III, testicular atrophy, occlusive azoospermia, etc.) that would impair participants response to treatment or has had known damage or injury to the vas deferens.
* Had any previous treatment with GnRH, gonadotropins (e.g., hCG, FSH) or androgens (e.g., testosterone, etc.). Note: Use of GnRH and gonadotropins for diagnostic testing purposes only is allowed. Participants with use of hCG and androgen therapy prior to the age of 2 years old can be included in the trial. Participants with transient use of androgens (i.e., for less than 2 weeks) that was stopped at least 6 months prior to signing informed consent can also be included in the trial.
* Has an untreated or inadequately treated pituitary or hypothalamic tumor.
* Have uncontrolled endocrinopathies, including thyroid, adrenal, and pituitary disorders not on stable replacement therapies.
* Has a history of active pituitary hypersecretion as evidenced by hyperprolactinemia or Cushing's disease, acromegaly, or any other active pituitary hypersecretion syndrome. (Note: Individuals who have been treated and are clinically stable, with no evidence of hypersecretion for at least 12 months prior to screening, may participate.
* Has had hypophysectomy within 12 months to the start of screening.
* Has history of oncologic chemotherapy treatment.
* Has had brain radiotherapy within 12 months of start of treatment for a primary tumor, or any history of brain radiotherapy for metastatic disease.
* Has diabetes mellitus.
* Has history of Human Immunodeficiency Virus (HIV).
* Has renal insufficiency, as determined by investigator, based on serum creatinine, blood urea nitrogen, and estimated glomerular filtration rate.
* Has clinically significant liver disease, including active viral hepatitis or cirrhosis. Individuals with a prior history of liver disease which is now inactive or successfully treated may be enrolled if all liver function values performed within the past year have been normal and within the normal range at Visit 1.
* Has had a recent history of recreational or illicit drug use, including marijuana; or routinely consumes >2 alcoholic drinks per day or >14 alcoholic drinks per week, or engages in binge drinking.
* Has an allergy/sensitivity to gonadotropins or its/their excipients.
* Has used an investigational drug and/or participated in any other clinical trial within the past 8 weeks (prior to Visit 2), or will participate in any other clinical trials (excluding surveys) during the course of this trial.

Ages: 14 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — All participants must be male.
Enrollment: 17 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2020-05-05 (Actual); Study Completion 2020-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (15):
- Brazil (3):
  - Centro de Diabetes Curitiba ( Site 0012), Curitiba
  - Hospital de Clinicas de Porto Alegre ( Site 0014), Porto Alegre
  - Hosp das Clinicas da Faculdade de Medicina da Univ de Sao Paulo ( Site 0015), São Paulo
- Rigshospitalet, University department of Growth and Reproduction ( Site 0051), Copenhagen, Denmark
- Italy (3):
  - AOU Careggi ( Site 0042), Florence
  - Policlinico Umberto I ( Site 0043), Roma
  - IRCCS Ospedale Pediatrico Bambino Gesu ( Site 0044), Roma
- Mexico (2):
  - Instituto Nacional de Pediatria ( Site 0007), Mexico City
  - Hospital Infantil de Mexico Federico Gomez ( Site 0006), Mexico City
- Russia (5):
  - Kazan State Medical University ( Site 0024), Kazan'
  - Federal State Budget Institution Endocrinological Research Center ( Site 0021), Moscow
  - City children polyclinic #44 ( Site 0025), Saint Petersburg
  - St.Petersburg State Pediatric Medical University ( Site 0023), Saint Petersburg
  - Republic Children Clinical Hospital ( Site 0022), Ufa
- Little Company of Mary Hospital ( Site 0017), Pretoria, South Africa

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Male participants with Hypogonadotropic Hypogonadism (HH) aged 14 to <18 years were enrolled in the study. A total of 17 participants were allocated to the study treatment arm.
Period: Overall Study
Arm/Group | Corifollitropin Alfa (CFA)+Human Chorionic Gonadotropin (hCG)
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Male participants with Hypogonadotropic Hypogonadism (HH) aged 14 to <18 years were enrolled in the study.
Arm/Group | Corifollitropin Alfa (CFA)+Human Chorionic Gonadotropin (hCG)
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.5 (0.9) [lower limit 0.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 1
  Unknown or Not Reported | 0
Testicular Volume (TV) [Mean (Standard Deviation); unit: mL] | 2.2 (1.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Log-Transformed Testicular Volume (TV) to Week 64
Description: Participants underwent testicular ultrasound of left and right testes at pre-specified time points to measure TV. TV was measured as the sum of volumes of left and right testes. The linear mixed model with a fixed effect for baseline and Week 64 and a random effect for participant was used to calculate the mean change in log-transformed TV and associated 95% confidence intervals (CIs) from baseline to Week 64. The geometric mean ratio and its 95% CIs for TV were obtained by exponentiation. The ratio > 1 indicated an increase in TV from baseline.
Time Frame: Baseline and Week 64
Population: All participants who received at least 1 dose of study treatment, who had a baseline and at least 1 post baseline TV value, had luteinizing hormone (LH) level ≤3 IU/L anytime in the study, had at least 12 weeks of Corifollitropin Alfa (CFA) and 24 weeks of CFA plus human chorionic gonadotropin (hCG) treatment, have last TV value within 4 weeks from last dose of CFA were analyzed.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Corifollitropin Alfa (CFA)+Human Chorionic Gonadotropin (hCG)
Number analyzed (Participants) | 13
mL
  Baseline | 1.5 (0.7)
  Week 64 | 14.5 (6.8)
Statistical Analysis 1: Comparison: Corifollitropin Alfa (CFA)+Human Chorionic Gonadotropin (hCG); Test type: Other — Linear Mixed Model; Geometric Mean Ratio = 9.43, 95% CI 2-sided [7.44 to 11.97]

2. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An adverse event was defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. The number of participants who experienced an AE was reported.
Time Frame: Up to approximately 71 Weeks
Population: All participants who received at least 1 dose of study treatment were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Corifollitropin Alfa (CFA)+Human Chorionic Gonadotropin (hCG)
Number analyzed (Participants) | 17
Participants | 16

3. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An adverse event was defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. The number of participants who discontinued study treatment due to an AE was reported.
Time Frame: Up to approximately 64 Weeks
Population: All participants who received at least 1 dose of study treatment were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Corifollitropin Alfa (CFA)+Human Chorionic Gonadotropin (hCG)
Number analyzed (Participants) | 17
Participants | 1

4. Primary Outcome: Percentage of Participants With Anti-Corifollitropin Alfa (CFA) Antibodies
Description: Blood samples were collected at pre-specified time points to assess anti-CFA antibodies. The percentage of participants with anti-CFA antibodies after administration of CFA were reported.
Time Frame: Up to approximately 71 Weeks
Population: All participants who received at least 1 dose of study treatment were analyzed.
Measure: Number; unit: Percentage of Participants
Arm/Group | Corifollitropin Alfa (CFA)+Human Chorionic Gonadotropin (hCG)
Number analyzed (Participants) | 17
Percentage of Participants | 0

5. Secondary Outcome: Change From Baseline in Serum Inhibin B Concentration to Week 64
Description: Serum Inhibin B concentration is a surrogate marker for spermatogenesis in males. Blood samples were collected at baseline and Week 64 post dose to report the mean change from baseline in serum inhibin concentration to Week 64. A mean change from baseline in serum inhibin B concentration to Week 64 was reported. A positive value indicated a higher serum inhibin concentration level.
Time Frame: Baseline and Week 64
Population: All participants who received at least 1 dose of study treatment who had a baseline and at least 1 post baseline TV value, had LH level ≤3 IU/L anytime in the study, had at least 12 weeks of CFA and 24 weeks of CFA plus hCG treatment, have last TV value within 4 weeks from last dose of CFA and had a baseline and at least 1 post baseline inhibin value were analyzed.
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Corifollitropin Alfa (CFA)+Human Chorionic Gonadotropin (hCG)
Number analyzed (Participants) | 13
ng/L
  Baseline | 31.92 (35.30) [lower limit 35.30]
  Baseline to Week 64 | 91.46 (59.25) [lower limit 59.25]

6. Secondary Outcome: Growth Velocity at Week 36
Description: Growth velocity is the rate of change in height measurement and is a marker for pubertal progress. Height was measured using a wall-mounted calibrated stadiometer. A mixed model was used to assess the overall growth velocity slope over the 36-week treatment period using the slopes estimated from an overall mixed random intercept and random slope model of height (cm) and time (yr) and age as covariates.
Time Frame: Week 36
Population: All participants who received at least 1 dose of study treatment, had a baseline and at least 1 post baseline TV value, had LH level ≤3 IU/L anytime in the study, had at least 12 weeks of CFA and 24 weeks of CFA plus hCG treatment, had last TV value within 4 weeks from last dose of CFA and had a baseline and post baseline height records at Week 36 were analyzed.
Measure: Least Squares Mean (Standard Error); unit: cm/year
Arm/Group | Corifollitropin Alfa (CFA)+Human Chorionic Gonadotropin (hCG)
Number analyzed (Participants) | 13
cm/year | 8.3 (1.1) [lower limit 1.1]

7. Secondary Outcome: Growth Velocity at Week 64
Description: Growth velocity is the rate of change in height measurement and is a marker for pubertal progress. Height was measured using a wall-mounted calibrated stadiometer. A mixed model was used to assess the overall growth velocity slope over the 64-week treatment period using the slopes estimated from an overall mixed random intercept and random slope model of height (cm) and time (year) and age as covariates.
Time Frame: Week 64
Population: All participants who received at least 1 dose of study treatment, had a baseline and at least 1 post baseline TV value, had LH level ≤3 IU/L anytime in the study, had at least 12 weeks of CFA and 24 weeks of CFA plus hCG treatment, had last TV value within 4 weeks from last dose of CFA and had a baseline and post baseline height records at Week 64 were analyzed.
Measure: Least Squares Mean (Standard Error); unit: cm/year
Arm/Group | Corifollitropin Alfa (CFA)+Human Chorionic Gonadotropin (hCG)
Number analyzed (Participants) | 12
cm/year | 7.6 (1.0) [lower limit 1.0]

8. Secondary Outcome: Change From Baseline in Tanner Stage (TS) of Pubertal Development for Pubic Hair to Week 12, Week 36, and Week 64
Description: Male participants were assessed clinically for pubertal development using the TS for pubic hair (range: Tanner I-V). TS describes sexual maturity stages (no better or worse outcome) as: Tanner I: prepubertal state, Tanner II: small amount of long, downy hair with slight pigmentation at the base of the penis and scrotum, Tanner III: hair becomes more coarse and curly, and begins to extend laterally, Tanner IV: adult-like hair quality, extending across pubis but sparing medial thighs and Tanner V: hair extends to medial surface of the thigh. The number of participants in each Tanner stage at baseline and categorical change from baseline in Tanner stages to Weeks 12, 36 and 64 were reported.
Time Frame: Baseline, Week 12, Week 36, and Week 64
Population: All participants who received at least 1 dose of study treatment who had a baseline and at least 1 post baseline TV value, had LH level ≤3 IU/L anytime in the study, had at least 12 weeks of CFA and 24 weeks of CFA plus hCG treatment, have last TV value within 4 weeks from last dose of CFA were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Corifollitropin Alfa (CFA)+Human Chorionic Gonadotropin (hCG)
Number analyzed (Participants) | 13
Participants
  Baseline (BL) Tanner I | 6
  BL Tanner II | 6
  BL Tanner III | 1
  BL Tanner IV | 0
  BL Tanner V | 0
  BL Tanner I to Week 12 Tanner I | 5
  BL Tanner I to Week 12 Tanner II | 1
  BL Tanner II to Week 12 Tanner II | 5
  BL Tanner II to Week 12 Tanner III | 1
  BL Tanner III to Week 12 Tanner III | 1
  BL Tanner I to Week 36 Tanner II | 2
  BL Tanner I to Week 36 Tanner III | 4
  BL Tanner II to Week 36 Tanner II | 2
  BL Tanner II to Week 36 Tanner III | 4
  BL Tanner III to Week 36 Tanner IV | 1
  BL Tanner I to Week 64 Tanner III | 3
  BL Tanner I to Week 64 Tanner IV | 1
  BL Tanner I to Week 64 Tanner V | 2
  BL Tanner II to Week 64 Tanner III | 1
  BL Tanner II to Week 64 Tanner IV | 3
  BL Tanner II to Week 64 Tanner V | 1
  BL Tanner II to Week 64 Unknown | 1
  BL Tanner III to Week 64 Tanner IV | 1

9. Secondary Outcome: Change From Baseline in TS of Pubertal Development for Genital Growth to Week 12, Week 36, and Week 64
Description: Male participants were assessed clinically for pubertal development using TS for genital growth (range: Tanner I-V). TS describes sexual maturity stages (no better or worse outcome) as: Tanner I: prepubertal (TV <1.5 ml; small penis), Tanner II: TV 1.6-6ml; skin on scrotum thins, reddens and enlarges; penis length unchanged, Tanner III: TV 6-12ml; scrotum enlarges further; penis begins to lengthen Tanner IV: TV 12-20ml; scrotum enlarges further and darkens; penis increases in length and circumference, and Tanner V: TV >20ml; adult scrotum and penis. The number of participants in each Tanner stage at baseline and categorical change from baseline in Tanner stages to Weeks 12, 36 and 64 were reported.
Time Frame: Baseline, Week 12, Week 36, and Week 64
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Corifollitropin Alfa (CFA)+Human Chorionic Gonadotropin (hCG)
Number analyzed (Participants) | 13
Participants
  Baseline (BL) Tanner I | 12
  BL Tanner II | 1
  BL Tanner III | 0
  BL Tanner IV | 0
  BL Tanner V | 0
  BL Tanner I to Week 12 Tanner I | 9
  BL Tanner I to Week 12 Tanner II | 3
  BL Tanner II to Week 12 Tanner II | 1
  BL Tanner I to Week 36 Tanner I | 2
  BL Tanner I to Week 36 Tanner II | 1
  BL Tanner I to Week 36 Tanner III | 8
  BL Tanner I to Week 36 Tanner IV | 1
  BL Tanner II to Week 36 Tanner II | 1
  BL Tanner I to Week 64 Tanner II | 1
  BL Tanner I to Week 64 Tanner III | 4
  BL Tanner I to Week 64 Tanner IV | 4
  BL Tanner I to Week 64 Tanner V | 2
  BL Tanner I to Week 64 Unknown | 1
  BL Tanner II to Week 64 Tanner III | 1

10. Secondary Outcome: Mean Serum Concentration of CFA
Description: Blood samples were collected at pre-specified time points (Day 1 (predose, 6-24 hours postdose after 1st dose), Day 3 (32-52 hours postdose after 1st dose), Day 5 (72-120 hours postdose after 1st dose), Day 8 (144-192 hours postdose after 1st dose), Day 11 (216-244 hours postdose after 1st dose), Day 29 (predose prior to 2nd dose; no hCG), Day 85 (predose, prior to 4th dose; no hCG), Day 169 (predose prior to 7th dose; with hCG co-administration), Day 253 (predose prior to 10th dose with hCG co-administration), Day 337 (predose prior to 13th dose; with hCG co-administration), Days 449 and 456 (postdose)) to report the mean serum concentration of CFA.
Time Frame: Day 1: predose, 6-24 hours postdose; Day 3: 32-52 hours postdose; Day 5: 72-120 hours postdose; Day 8: 144-192 hours postdose; Day 11: 216-244 hours postdose; Days 29, 85, 169, 253, 337: predose; Days 449, 456: postdose
Population: All enrolled participants in the study were analyzed.
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Corifollitropin Alfa (CFA)+Human Chorionic Gonadotropin (hCG)
Number analyzed (Participants) | 17
ng/L
  Predose Day 1: number analyzed (Participants) | 16
  Predose Day 1 | 0.0 (0.0)
  Postdose Day 1 (6-24 hours): number analyzed (Participants) | 16
  Postdose Day 1 (6-24 hours) | 4100 (2630)
  Postdose Day 3 (32-52 hours) | 5880 (1640)
  Postdose Day 5 (72-120 hours) | 4240 (1180)
  Postdose Day 8 (144-192 hours): number analyzed (Participants) | 16
  Postdose Day 8 (144-192 hours) | 2110 (864)
  Postdose Day 11 (216-264 hours) | 1150 (655)
  Predose Day 29: number analyzed (Participants) | 16
  Predose Day 29 | 480 (348)
  Predose Day 85 | 695 (1310)
  Predose Day 169 | 691 (1060)
  Predose Day 253 | 301 (297)
  Predose Day 337: number analyzed (Participants) | 16
  Predose Day 337 | 556 (1260)
  Postdose Day 449: number analyzed (Participants) | 16
  Postdose Day 449 | 864 (1290)
  Postdose Day 456: number analyzed (Participants) | 16
  Postdose Day 456 | 0.0 (0.0)

11. Secondary Outcome: Change From Baseline in Testicular Echogenicity to Week 12, Week 36, and Week 64
Description: Testicular Echogenicity was determined by evaluating the sonographic patterns obtained on testicular ultrasound of right and left testes at baseline, Week 12, Week 36 and 64. The sonographic patterns were assessed by central imaging unit by an independent radiologist and categorized as Hypoechoic (decreased echogenicity as compared to echogenicity at baseline), Isoechoic (same echogenicity as compared to echogenicity at baseline) and Hyperechoic (increased echogenicity as compared to echogenicity at baseline). The number of participants with a sonographic pattern at Weeks 12, 36 and 64 were reported.
Time Frame: Baseline, Week 12, Week 36, and Week 64
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Corifollitropin Alfa (CFA)+Human Chorionic Gonadotropin (hCG)
Number analyzed (Participants) | 13
Participants
  Left Testes: Baseline (BL) to Week 12: Hypoechoic | 2
  Left Testes: BL to Week 12: Isoechoic | 10
  Left Testes: BL to Week 12: Hyperechoic | 1
  Right Testes: BL to Week 12: Hypoechoic | 1
  Right Testes: BL to Week 12: Isoechoic | 12
  Left Testes: BL to Week 36: Hypoechoic | 2
  Left Testes: BL to Week 36: Isoechoic | 10
  Left Testes: BL to Week 36: Hyperechoic | 1
  Right Testes: BL to Week 36: Hypoechoic | 1
  Right Testes: BL to Week 36: Isoechoic | 9
  Right Testes: BL to Week 36: Hyperechoic | 3
  Left Testes: BL to Week 64: Hypoechoic | 2
  Left Testes: BL to Week 64: Isoechoic | 8
  Left Testes: BL to Week 64: Hyperechoic | 3
  Right Testes: BL to Week 64: Isoechoic | 10
  Right Testes: BL to Week 64: Hyperechoic | 3

12. Secondary Outcome: Change From Baseline in Luteinizing Hormone (LH) to Week 12, Week 36, and Week 64
Description: LH is a gonadotropin secreted from the anterior pituitary and is a marker for spontaneous puberty. Blood samples were collected at baseline, Week 12, Week 36 and Week 64 to report the mean change from baseline in LH level to Weeks 12, 36 and 64.
Time Frame: Baseline, Week 12, Week 36, and Week 64
Population: All participants who received at least 1 dose of study treatment who had a baseline and at least 1 post baseline TV value, had LH level ≤3 IU/L anytime in the study, had at least 12 weeks of CFA and 24 weeks of CFA plus hCG treatment, had last TV value within 4 weeks from last dose of CFA and had a baseline and post baseline LH values at Weeks 12, 36 and 64 were analyzed.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Corifollitropin Alfa (CFA)+Human Chorionic Gonadotropin (hCG)
Number analyzed (Participants) | 13
IU/L
  Baseline | 0.25 (0.24)
  Baseline to Week 12 | -0.08 (0.15)
  Baseline to Week 36: number analyzed (Participants) | 12
  Baseline to Week 36 | -0.13 (0.25)
  Baseline to Week 64 | -0.14 (0.25)

13. Secondary Outcome: Change From Baseline in Calculated Free Testosterone (T) to Week 12, Week 36, and Week 64
Description: Blood samples were collected at baseline, Week 12, Week 36 and Week 64 to report the mean change from baseline in T level to Weeks 12, 36 and 64. The change from baseline in T level to Week 12, 36, and 64 could not be calculated as planned because only 2 participants had baseline T level values which were insufficient to provide the trend change from baseline in T level to Week 12, 36, and 64.
Time Frame: Baseline, Week 12, Week 36, and Week 64
Population: All participants who received at least 1 dose of study treatment who had a baseline and at least 1 post baseline TV value, had LH level ≤3 IU/L anytime in the study, had at least 12 weeks of CFA and 24 weeks of CFA + hCG treatment, had last TV value within 4 weeks from last CFA dose and had a baseline and post baseline T value at Week 12, 36 and 64 were to be analyzed.
Arm/Group | Corifollitropin Alfa (CFA)+Human Chorionic Gonadotropin (hCG)
Number analyzed (Participants) | 0

14. Secondary Outcome: Change From Baseline in Total Testosterone (Total T) to Week 12, Week 36, and Week 64
Description: Total T is a marker for progress of puberty in males. Total T levels increase during puberty as the testes respond to the gonadotropins. Blood samples were collected at baseline, Week 12, Week 36 and Week 64 post dose to report the mean change from baseline in Total T level to Weeks 12, 36 and 64. A negative value indicated a lower Total T level.
Time Frame: Baseline, Week 12, Week 36, and Week 64
Population: All participants who received at least 1 dose of study treatment who had a baseline and at least 1 post baseline TV value, had LH level ≤3 IU/L anytime in the study, had at least 12 weeks of CFA and 24 weeks of CFA plus hCG treatment, had last TV value within 4 weeks from last dose of CFA and had a baseline and post baseline Total T value at Week 12, 36 and 64 were analyzed.
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Corifollitropin Alfa (CFA)+Human Chorionic Gonadotropin (hCG)
Number analyzed (Participants) | 13
ug/L
  Baseline | 0.11 (0.12)
  Baseline to Week 12: number analyzed (Participants) | 12
  Baseline to Week 12 | -0.01 (0.07)
  Baseline to Week 36 | 4.87 (3.97)
  Baseline to Week 64 | 5.31 (3.31)

15. Secondary Outcome: Change From Baseline in Estradiol (E2) to Week 12, Week 36, and Week 64
Description: E2 levels rise during puberty in males when some of the T secreted is aromatized. Blood samples were collected at baseline, Week 12, Week 36 and Week 64 to report the mean change from baseline in E2 level to Weeks 12, 36 and 64. A positive value indicated a higher E2 level.
Time Frame: Baseline, Week 12, Week 36, and Week 64
Population: All participants who received at least 1 dose of study treatment who had a baseline and at least 1 post baseline TV value, had LH level ≤3 IU/L anytime in the study, had at least 12 weeks of CFA and 24 weeks of CFA plus hCG treatment, had last TV value within 4 weeks from last dose of CFA and had a baseline and post baseline E2 value at Week 12, 36 and 64 were analyzed.
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Corifollitropin Alfa (CFA)+Human Chorionic Gonadotropin (hCG)
Number analyzed (Participants) | 13
ng/L
  Baseline | 9.51 (0.00) [lower limit 0.00]
  Baseline to Week 12 | 0.81 (2.90) [lower limit 2.90]
  Baseline to Week 36 | 37.57 (28.73) [lower limit 28.73]
  Baseline to Week 64 | 45.58 (41.09) [lower limit 41.09]

16. Secondary Outcome: Change From Baseline in Sex Hormone-Binding Globulin (SHBG) to Week 12, Week 36, and Week 64
Description: SHBG is a blood protein that controls the amount of T body tissues in males. SHBG is regulated by the ratio of T and E2 levels in addition to other factors (thyroid hormone status, dietary factors, certain diseases and medications). Blood samples were collected at baseline, Week 12, Week 36 and Week 64 to report the mean change from baseline in SHBG level to Weeks 12, 36 and 64. A negative value indicated a lower SHBG level.
Time Frame: Baseline, Week 12, Week 36, and Week 64
Population: All participants who received at least 1 dose of study treatment who had a baseline and at least 1 post baseline TV value, had LH level ≤3 IU/L anytime in the study, had at least 12 weeks of CFA and 24 weeks of CFA plus hCG treatment, had last TV value within 4 weeks from last dose of CFA and had a baseline and post baseline SHBG value at Week 12, 36 and 64 were analyzed.
Measure: Mean (Standard Deviation); unit: ug/dL
Arm/Group | Corifollitropin Alfa (CFA)+Human Chorionic Gonadotropin (hCG)
Number analyzed (Participants) | 13
ug/dL
  Baseline | 1.53 (0.91)
  Baseline to Week 12 | 0.04 (0.45)
  Baseline to Week 36: number analyzed (Participants) | 12
  Baseline to Week 36 | -0.53 (0.73)
  Baseline to Week 64 | -0.68 (0.76)

17. Secondary Outcome: Change From Baseline in Anti-Müllerian Hormone (AMH) to Week 12, Week 36, and Week 64
Description: AMH is a marker for progress of puberty in males. Blood samples were collected at baseline, Week 12, Week 36 and Week 64 to report the mean change from baseline in AMH level to Weeks 12, 36 and 64. A negative value indicated a lower AMH level.
Time Frame: Baseline, Week 12, Week 36, and Week 64
Population: All participants who received at least 1 dose of study treatment who had a baseline and at least 1 post baseline TV value, had LH level ≤3 IU/L anytime in the study, had at least 12 weeks of CFA and 24 weeks of CFA plus hCG treatment, had last TV value within 4 weeks from last dose of CFA and had a baseline and post baseline AMH value at Week 12, 36 and 64 were analyzed.
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Corifollitropin Alfa (CFA)+Human Chorionic Gonadotropin (hCG)
Number analyzed (Participants) | 13
ug/L
  Baseline | 23.62 (11.07)
  Baseline to Week 12 | 17.98 (8.39)
  Baseline to Week 36: number analyzed (Participants) | 12
  Baseline to Week 36 | -10.23 (15.69)
  Baseline to Week 64 | -15.83 (11.58)

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious and non-serious AEs were collected for up to approximately 71 Weeks
Description: All participants who received at least one dose of study treatment were analyzed.
Arm/Group | Corifollitropin Alfa (CFA)+Human Chorionic Gonadotropin (hCG)
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 1/17
Other Adverse Events (participants affected / at risk) | 16/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Corifollitropin Alfa (CFA)+Human Chorionic Gonadotropin (hCG) (N=17)
Craniopharyngioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Corifollitropin Alfa (CFA)+Human Chorionic Gonadotropin (hCG) (N=17)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Gingival oedema (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3)
Injection site pain (General disorders) | 1 (2)
Oedema peripheral (General disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2)
Respiratory tract infection (Infections and infestations) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Tinea infection (Infections and infestations) | 1 (1)
Tracheitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Blood prolactin increased (Investigations) | 1 (1)
Blood testosterone decreased (Investigations) | 2 (2)
Blood testosterone free increased (Investigations) | 2 (2)
Blood testosterone increased (Investigations) | 4 (4)
Human chorionic gonadotropin increased (Investigations) | 1 (1)
Oestradiol increased (Investigations) | 5 (5)
Testicular scan abnormal (Investigations) | 1 (1)
Ultrasound testes abnormal (Investigations) | 1 (1)
Hyperphagia (Metabolism and nutrition disorders) | 1 (1)
Metabolic syndrome (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Cerebrovascular disorder (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 4 (4)
Migraine (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Pruritus genital (Reproductive system and breast disorders) | 1 (1)
Scrotal disorder (Reproductive system and breast disorders) | 1 (1)
Spermatocele (Reproductive system and breast disorders) | 5 (6)
Varicocele (Reproductive system and breast disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Acanthosis nigricans (Skin and subcutaneous tissue disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Hot flush (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-24): https://cdn.clinicaltrials.gov/large-docs/75/NCT03019575/Prot_SAP_000.pdf